CLINICAL TRIAL: NCT04767243
Title: Regenerative Potential of Advanced Platelet Rich Fibrin (A-PRF) and Bioactive Glass (Perioglas®) Bone Graft in the Treatment of Intrabony Defects; A Comparative Clinico Radiographic Study.
Brief Title: Regenerative Potential of Advanced Platelet Rich Fibrin and Bioactive Glass (Perioglas®).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, DR SURINDER SACHDEVA, PROFESSOR, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1597
Record Dates: First submitted 2021-02-09; First posted 2021-02-23 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Chronic Periodontitis; Bone Loss; Intrabony Periodontal Defect
Keywords: intrabony periodontal defect; regeneration; platelet rich fibrin; bioactive glass
MeSH Terms: conditions — Chronic Periodontitis; Bone Diseases, Metabolic | interventions — Bioglass

STUDY DESIGN:
Intervention Model Description: 45 sites with vertical intrabony alveolar defects will be selected. These defect sites will be allocated randomly into 3 groups as Group I, Group II and Group III.
  * Group I will be treated with open flap debridement and filled with A-PRF
  * Group II will be treated with open flap debridement and filled with Bioactive glass (Perioglas®)
  * Group III will be treated with open flap debridement and filled Bioactive glass (Perioglas®) and A-PRF.
Who Masked: Participant, Outcomes Assessor
Masking Description: patient and statistician will be masked about the treatment regimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- open flap debridement and filled with A-PRF (Sham Comparator): After phase 1 therapy, surgical procedure would be carried out in the selected patients under aseptic conditions. Full thickness mucoperiosteal Kirkland flap would be raised on both buccal and lingual sides using periosteal elevator. Pocket lining epithelium would be removed and a thorough debridement and root planing would be done in the intrabony defect by using Gracey curettes and universal curettes. After placement of A-PRF in bony defect site the mucoperiosteal flaps would be sutured for complete soft tissue closure.
  Interventions: Procedure: open flap debridement and filled with A-PRF ( Advanced platelet rich fibrin)
- open flap debridement and filled with Bioactive glass (Perioglas®) (Active Comparator): After phase 1 therapy, surgical procedure would be carried out in the selected patients under aseptic conditions. Full thickness mucoperiosteal Kirkland flap would be raised on both buccal and lingual sides using periosteal elevator. Pocket lining epithelium would be removed and a thorough debridement and root planing would be done in the intrabony defect by using Gracey curettes and universal curettes. After placement of Bioactive glass (Perioglas®) in bony defect site the mucoperiosteal flaps would be sutured for complete soft tissue closure.
  Interventions: Procedure: open flap debridement and filled with Bioactive glass (Perioglas®)
- with open flap debridement and filled Bioactive glass (Perioglas®) and A-PRF. (Active Comparator): After phase 1 therapy, surgical procedure would be carried out in the selected patients under aseptic conditions. Full thickness mucoperiosteal Kirkland flap would be raised on both buccal and lingual sides using periosteal elevator. Pocket lining epithelium would be removed and a thorough debridement and root planing would be done in the intrabony defect by using Gracey curettes and universal curettes. After placement of Bioactive glass (Perioglas®) along with A-PRF in bony defect site the mucoperiosteal flaps would be sutured for complete soft tissue closure.
  Interventions: Drug: open flap debridement and filled Bioactive glass (Perioglas®) and A-PRF

INTERVENTIONS:
Procedure: open flap debridement and filled with A-PRF ( Advanced platelet rich fibrin) — After phase 1 therapy, surgical procedure would be carried out in the selected patients under aseptic conditions. Full thickness mucoperiosteal Kirkland flap would be raised on both buccal and lingual sides using periosteal elevator. Pocket lining epithelium would be removed and a thorough debridement and root planing would be done in the intrabony defect by using Gracey curettes and universal curettes. After placement of A-PRF in bony defect site the mucoperiosteal flaps would be sutured for complete soft tissue closure.
  Arms: open flap debridement and filled with A-PRF
Procedure: open flap debridement and filled with Bioactive glass (Perioglas®) — After phase 1 therapy, surgical procedure would be carried out in the selected patients under aseptic conditions. Full thickness mucoperiosteal Kirkland flap would be raised on both buccal and lingual sides using periosteal elevator. Pocket lining epithelium would be removed and a thorough debridement and root planing would be done in the intrabony defect by using Gracey curettes and universal curettes. After placement of perioglas in bony defect site the mucoperiosteal flaps would be sutured for complete soft tissue closure.
  Other Names: perioglas
  Arms: open flap debridement and filled with Bioactive glass (Perioglas®)
Drug: open flap debridement and filled Bioactive glass (Perioglas®) and A-PRF — After phase 1 therapy, surgical procedure would be carried out in the selected patients under aseptic conditions. Full thickness mucoperiosteal Kirkland flap would be raised on both buccal and lingual sides using periosteal elevator. Pocket lining epithelium would be removed and a thorough debridement and root planing would be done in the intrabony defect by using Gracey curettes and universal curettes. After placement of perioglas with A-PRF in bony defect site the mucoperiosteal flaps would be sutured for complete soft tissue closure.
  Other Names: perioglas
  Arms: with open flap debridement and filled Bioactive glass (Perioglas®) and A-PRF.

SUMMARY:
The aim of this study is to evaluate and compare the regenerative potential of Advanced Platelet Rich Fibrin (A-PRF) and Bioactive Glass (Perioglas®) bone graft in the treatment of intrabony defects in chronic periodontitis patients.

DETAILED DESCRIPTION:
45 sites with vertical intrabony alveolar defects will be selected. These defect sites will be allocated randomly into 3 groups as Group I, Group II and Group III.

* Group I will be treated with open flap debridement and filled with A-PRF
* Group II will be treated with open flap debridement and filled with Bioactive glass (Perioglas®)
* Group III will be treated with open flap debridement and filled Bioactive glass (Perioglas®) and A-PRF.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 to 55 years.
* Gender: Both males and females will be included in the study.
* Co-operative and motivated patients committed to oral hygiene.
* Patients exhibiting intrabony defects.

Exclusion Criteria:

* Patients with contraindication to periodontal surgery & local anesthesia.
* Any systemic disease affecting the bone density and outcome of periodontal therapy.
* Smokers, alcoholics, and patients with other adverse habits.
* Pregnant, nursing and menopausal women.
* Any known allergy/ hypersensitivity to any product used in this study.
* Patients on long-term systemic therapy (antibiotics, anti-inflammatory bisphosphonates, hormonal replacement therapy and any other), taking any drug known to have periodontal implications that may interfere with wound healing.
* Patients taking any anti-platelet and anticoagulant medication.
* Patients who have undergone periodontal treatment within a period of past 1 year.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
probing depth | baseline, 3 months, 6 months
  change in probing pocket depth
relative attachment level | baseline, 3 months, 6 months
  change in attachment level
radiographic linear bone change | change from baseline to 6 months
  radiographic linear bone change through radiographic grid

SECONDARY OUTCOMES:
Plaque index site specific | baseline, 3 months, 6 months
  Plaque index -Silness and Loe
Gingival index site specific | baseline, 3 months, 6 months
  Gingival index- Loe and Silness

CONTACTS AND LOCATIONS:
Overall Officials: surinder sachdeva, M.D.S., Principal Investigator — PROFESSOR
Locations (1):
- Department of Periodontology, M.M. College of Dental Sciences and Research., Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghanaati S, Booms P, Orlowska A, Kubesch A, Lorenz J, Rutkowski J, Landes C, Sader R, Kirkpatrick C, Choukroun J. Advanced platelet-rich fibrin: a new concept for cell-based tissue engineering by means of inflammatory cells. J Oral Implantol. 2014 Dec;40(6):679-89. doi: 10.1563/aaid-joi-D-14-00138. PMID 24945603
- [Background] Mengel R, Schreiber D, Flores-de-Jacoby L. Bioabsorbable membrane and bioactive glass in the treatment of intrabony defects in patients with generalized aggressive periodontitis: results of a 5-year clinical and radiological study. J Periodontol. 2006 Oct;77(10):1781-7. doi: 10.1902/jop.2006.060029. PMID 17032123